CLINICAL TRIAL: NCT06536348
Title: PARKINSON BRASIL - Database on Motor and Non-Motor Aspects of Parkinson's Disease in Brazil
Status: Not yet recruiting | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Núcleo de Inovação e Avaliação Tecnológica em Saúde (Unknown); Ambulatório de Doença de Parkinson e Distúrbios do Movimento do Hospital de Clínicas de Uberlândia (Unknown); Associação Parkinson Goiás (Unknown); Centro Universitário Araguaia (UniAraguaia) (Unknown); Laboratório de Análise de Movimento e Processamento de Sinais (Unknown)
Responsible Party: Principal Investigator, Adriano de Oliveira Andrade, Professor, Federal University of Uberlandia
Other Study IDs: 81274724.0.0000.5152; 13585 (Other: Empresa Brasileira de Serviços Hospitalares (EBSERH))
Record Dates: First submitted 2024-07-28; First posted 2024-08-02 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; motor assessment; non-motor assessment; database; computer vision; inertial sensors
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: Group of subjects with Parkinson's disease
- Control group: Neurological healthy subjects

SUMMARY:
This is an observational, cross-sectional study with a control group, with the general objective of developing and evaluating a national database, unprecedented in Brazil, containing clinical, epidemiological, motor, and non-motor aspects of Parkinson's disease (PD). The database will be open and accessible to national and international researchers in order to contribute to the advancement of research related to PD. The aim is to collect data, in a paired way, from a control group and an experimental group. Data collection will include the application of questionnaires, the execution of motor activities, and clinical scales. Information that can identify the participants will be removed from the database for later storage in a repository. Quantitative, qualitative, and descriptive variables from the database will be estimated in order to characterise and contrast the groups studied. The results of this study will contribute to a better characterization of the staging of PD as a function of the epidemiological, motor, and non-motor aspects evaluated, as well as to the development of technologies and methods that can be applied in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group: (i) present a neurological diagnosis of Parkinson's disease; (ii) be classified between stages I to IV of the Hoehn & Yahr Scale; (iii) have central visual acuity equal to or greater than 20/40 (equivalent to 0.50) in each eye or equal to or greater than 20/30 (equivalent to 0.66) in one eye according to the Snellen scale.
* Control group: (i) not having a neurological diagnosis of Parkinson's disease or other neurological disease that resembles PD; (ii) have central visual acuity equal to or greater than 20/40 (equivalent to 0.50) in each eye or equal to or greater than 20/30 (equivalent to 0.66) in one eye according to the Snellen scale.

Exclusion Criteria:

For both groups, individuals who have other neurological or musculoskeletal diseases that interfere with the execution of the tests will be excluded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Experimental group: Individuals diagnosed with Parkinson's disease
  * Control group: Individuals not having Parkinson's disease (PD) or other neurological disease that resembles PD;
Sampling Method: Non-Probability Sample
Enrollment: 958 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2034-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Sex | 10 years
  Sex: male, female
Age | 10 years
  Age in years
Length of schooling | 10 years
  Length of schooling in years
Weight | 10 years
  Weight in kg
Height | 10 years
  Height in cm
Blood type | 10 years
  Blood type: A+, A-, B+, B-, O+, O-, AB+, AB-
Economic Rating Score | 10 years
  Economic rating as given by the Brazilian Economic Classification Criteria (Brazilian Criteria) - https://www.abep.org/criterioBr/01_cceb_2022_eng.pdf
Primary ICD | 10 years
  Primary disorder classification according to the International Statistical Classification of Diseases and Related Health Problems (ICD) https://www.who.int/standards/classifications/classification-of-diseases
Secondary ICDs | 10 years
  Secondary disorder according to the International Statistical Classification of Diseases and Related Health Problems (ICD) https://www.who.int/standards/classifications/classification-of-diseases
Medications in use | 10 years
  name and daily dose of medications
Family history related to the primary ICD | 10 years
  Is there family history related to the primary ICD? (yes, no)
Date of symptom onset related to the primary ICD | 10 years
  date
Date of diagnosis related to the primary ICD | 10 years
  date
Current city of residence | 10 years
  City of residence in Brazil
Current state of residence | 10 years
  State of residence in Brazil
Civil status | 10 years
  married, single, divorced, and widowed
Housing classification | 10 years
  Housing classification by type of housing ownership rights: State-owned housing, Municipality-owned housing, Natural person's owned housing, Legal person's owned housing, Private renting, Other
Household size | 10 years
  The number of adults and children living in a home
Laterality | 10 years
  Laterality refers to the preference for using one side of the body over the other and is most commonly associated with hand dominance, such as being right-handed or left-handed, e.g., Right-handedness, Left-handedness, Ambidexterity, Mixed-handedness (Cross-dominance).
Use of technology | 10 years
  Verification if the participant has had contact with one of the following devices: mobile, personal computer, mouse, webcam, keyboard, microphone, earphone.
Occupation | 10 years
  Profession according to the Brazilian Classification of Occupation (https://www.mtecbo.gov.br/cbosite/pages/home.jsf)
Monthly wage | 10 years
  Monthly wage in Brazilian Reais
Head movement amplitude | 10 years
  Head movement amplitude in degrees
Head movement speed | 10 years
  Head movement speed in degrees per second
Facial expression | 10 years
  Facial expression evaluation according to the Facial Action Coding System (FACS)
Saccadic eye movement | 10 years
  Speed and regularity of eye movement (degrees per second and latency in ms)
Smooth pursuit eye movement | 10 years
  Smooth pursuit are quantified by the gain (how well the eyes follow the target in speed) and phase (distance to the target during pursuit)
Handwriting movement analysis | 10 years
  Handwriting speed (seconds) and quality
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 10 years
  Clinical scale for measuring signs and symptoms of Parkinson's disease (https://www.movementdisorders.org/MDS/MDS-Rating-Scales/MDS-Unified-Parkinsons-Disease-Rating-Scale-MDS-UPDRS.htm?gad_source=1&gclid=CjwKCAjwnqK1BhBvEiwAi7o0X6DuHrFh3qftNQ1N9AGWMkFo4BpG6b3hAFWnoh2Dwu86DPY53ZXpKRoCBRYQAvD_BwE)
  Each item of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale will be evaluated as 0: Normal; 1: Slight; 2: Mild; 3: Moderate; 4: Severe.
  The minimum value of the scale is 0, whereas the maximum value is 4. Higher scores mean a worse outcome.
Depression | 10 years
  Depression measured according to the Geriatric Depression Scale (GDS) https://geriatrictoolkit.missouri.edu/cog/GDS_SHORT_FORM.PDF
  The Geriatric Depression Scale has 15 items. The minimum total score is zero, and the maximum is 15. Higher scores mean a worse outcome.
Visual Acuity | 10 years
  Visual Acuity measured according to the Snellen test (https://www.ncbi.nlm.nih.gov/books/NBK558961/)
Cognition | 10 years
  Cognition measured according to the Montreal Cognitive Assessment (MOCA) scale
  The Montreal Cognitive Assessment (MoCA) is a 30-point test. The minimum total score is zero, and the maximum is 30. Higher scores mean a better outcome.
Dysarthria | 10 years
  Dysarthria measured according to the protocol for the evaluation of central dysartries in patients with Parkinson's Disease (https://doi.org/10.1590/S1516-18462011005000030)
Hand movement | 10 years
  Hand movement in degrees per second

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Andrade, PhD, Principal Investigator — Federal University of Uberlandia
Locations (5):
- Brazil (5):
  - Laboratório de Análise de Movimento e Processamento de Sinais, Brasília, Federal District
  - Centro Universitário Araguaia (UniAraguaia), Goiânia, Goiás
  - Associação Parkinson Goiás, Goiânia, Goiás
  - Ambulatório de Doença de Parkinson e Distúrbios do Movimento do Hospital de Clínicas de Uberlândia, Uberlândia, Minas Gerais
  - Núcleo de Inovação e Avaliação Tecnológica em Saúde / Centre for Innovation and Technology Assessment in Health, Uberlândia, Minas Gerais

IPD SHARING:
Plan to Share IPD: Yes
The data will be anonymised, stored in a safe and international plataform (Zenodo - https://github.com/NIATS-UFU). Only information that can be used to identify the subjects will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Researchers that wish to have access to the data can request access at https://github.com/NIATS-UFU. Full access will be granted for research purposes.

REFERENCES:
- [Background] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Background] World Health Organization, Parkinson disease, 2023.
- [Background] Barbosa MT, Caramelli P, Maia DP, Cunningham MC, Guerra HL, Lima-Costa MF, Cardoso F. Parkinsonism and Parkinson's disease in the elderly: a community-based survey in Brazil (the Bambui study). Mov Disord. 2006 Jun;21(6):800-8. doi: 10.1002/mds.20806. PMID 16482566
- [Background] Vale TC, Barbosa MT, Resende EPF, Maia DP, Cunningham MCQ, Guimaraes HC, Machado JCB, Teixeira AL, Cardoso F, Caramelli P. Parkinsonism in a population-based study of individuals aged 75+ years: The Pieta study. Parkinsonism Relat Disord. 2018 Nov;56:76-81. doi: 10.1016/j.parkreldis.2018.06.030. Epub 2018 Jun 19. PMID 29934195
- [Background] Simon DK, Tanner CM, Brundin P. Parkinson Disease Epidemiology, Pathology, Genetics, and Pathophysiology. Clin Geriatr Med. 2020 Feb;36(1):1-12. doi: 10.1016/j.cger.2019.08.002. Epub 2019 Aug 24. PMID 31733690
- [Background] Obeso JA, Rodriguez-Oroz MC, Rodriguez M, Lanciego JL, Artieda J, Gonzalo N, Olanow CW. Pathophysiology of the basal ganglia in Parkinson's disease. Trends Neurosci. 2000 Oct;23(10 Suppl):S8-19. doi: 10.1016/s1471-1931(00)00028-8. PMID 11052215
- [Background] Tysnes OB, Storstein A. Epidemiology of Parkinson's disease. J Neural Transm (Vienna). 2017 Aug;124(8):901-905. doi: 10.1007/s00702-017-1686-y. Epub 2017 Feb 1. PMID 28150045
- [Background] Dickson JM, Grunewald RA. Somatic symptom progression in idiopathic Parkinson's disease. Parkinsonism Relat Disord. 2004 Dec;10(8):487-92. doi: 10.1016/j.parkreldis.2004.05.005. PMID 15542009
- [Background] Cabral AM, Lora-Millan JS, Pereira AA, Rocon E, Andrade AO. On the Effect of Vibrotactile Stimulation in Essential Tremor. Healthcare (Basel). 2024 Feb 9;12(4):448. doi: 10.3390/healthcare12040448. PMID 38391822
- [Background] Cardoso Mendes L, Abreu Rosa de Sa A, Alves Marques I, Morere Y, de Oliveira Andrade A. RehaBEElitation: the architecture and organization of a serious game to evaluate motor signs in Parkinson's disease. PeerJ Comput Sci. 2023 Mar 15;9:e1267. doi: 10.7717/peerj-cs.1267. eCollection 2023. PMID 37346638
- [Background] S. Costa, I. A. Marques, A. Bevilaqua, A. Rabelo, L. Luiz, A. Cabral, N. Faustino, M. Okereke, M. Fraga Vieira e A. de Oliveira Andrade, "Biomechanical Evaluation of an Exoskeleton for Rehabilitation of Individuals with Parkinson's Disease," IRBM, vol. 44, p. 100741, February 2023
- [Background] L. C. Mendes, A. M. Cabral, C. M. Alves, Y. Morère e A. de Oliveira Andrade, "Objective assessment of tremor in Parkinson's disease using the RehaBEElitation serious game," em 2023 IEEE International Conference on Metrology for eXtended Reality, Artificial Intelligence and Neural Engineering (MetroXRAINE), 2023
- [Background] Mendes LC, Marques IA, Alves CM, Vieira MF, Junior EAL, Pereira AA, Naves ELM, Oliveira FHM, Bourhis G, Pino P, Morere Y, Andrade AO. Multidimensional Assessment of Individuals with Parkinson's Disease: Development and Structure Validation of a Self-Assessment Questionnaire. Healthcare (Basel). 2022 Sep 21;10(10):1823. doi: 10.3390/healthcare10101823. PMID 36292272
- [Background] Nobrega LR, Rocon E, Pereira AA, Andrade AO. A Novel Physical Mobility Task to Assess Freezers in Parkinson's Disease. Healthcare (Basel). 2023 Jan 31;11(3):409. doi: 10.3390/healthcare11030409. PMID 36766984
- [Background] L. C. Mendes, A. Moura Cabral, C. M. Alves, Y. Morere, I. A. Marques e A. de Oliveira Andrade, "Objective Evaluation of Bradykinesia Using the RehaBEElitation Serious Game," em 2022 IEEE Workshop on Complexity in Engineering (COMPENG), 2022.
- [Background] Machado AR, Zaidan HC, Paixao AP, Cavalheiro GL, Oliveira FH, Junior JA, Naves K, Pereira AA, Pereira JM, Pouratian N, Zhuo X, O'Keeffe A, Sharim J, Bordelon Y, Yang L, Vieira MF, Andrade AO. Feature visualization and classification for the discrimination between individuals with Parkinson's disease under levodopa and DBS treatments. Biomed Eng Online. 2016 Dec 30;15(1):169. doi: 10.1186/s12938-016-0290-y. PMID 28038673
- [Background] Rabelo AG, Neves LP, Paixao APS, Oliveira FHM, de Souza LAPS, Vieira MF, Pereira AA, Andrade AO. Objective Assessment of Bradykinesia Estimated from the Wrist Extension in Older Adults and Patients with Parkinson's Disease. Ann Biomed Eng. 2017 Nov;45(11):2614-2625. doi: 10.1007/s10439-017-1908-3. Epub 2017 Aug 29. PMID 28852889
- [Background] L. C. V. Ferreira, A. G. Rabelo, M. F. Vieira, A. A. Pereira e A. d. O. Andrade, "Gait variability and symmetry assessment with inertial sensors for quantitative discrimination of Trendelenburg sign in total hip arthroplasty patients: a pilot study based on convenience sampling," Research on Biomedical Engineering, vol. 34, p. 65-72, March 2018.
- [Background] Oliveira FHM, Machado ARP, Andrade AO. On the Use of t-Distributed Stochastic Neighbor Embedding for Data Visualization and Classification of Individuals with Parkinson's Disease. Comput Math Methods Med. 2018 Nov 4;2018:8019232. doi: 10.1155/2018/8019232. eCollection 2018. PMID 30532798
- [Background] National Commission for the Incorporation of Technologies in the SUS - CONITEC, Clinical Protocol and Therapeutic Guidelines Parkinson's Disease, 2017.
- [Background] A. S. Fracassi, A. R. Gatto, S. Weber, A. A. Spadotto, P. W. Ribeiro and A. O. Schelp,
- [Background] Woo EH, White P, Lai CW. Ergonomics standards and guidelines for computer workstation design and the impact on users' health - a review. Ergonomics. 2016 Mar;59(3):464-75. doi: 10.1080/00140139.2015.1076528. Epub 2015 Sep 24. PMID 26224145
- [Background] J. F. Cecato, J. M. Montiel, D. Bartholomeu and J. E. Martinelli,